CLINICAL TRIAL: NCT05661500
Title: The Effect of Creative Drama Method on Nursing Students' Knowledge and Skills Regarding Postmortem Care
Brief Title: The Effect of Creative Drama on Postmortem Care in Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Lutfiye Nur Uzun, PhD Student, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AIBU-HEM-UZUN-001
Record Dates: First submitted 2022-12-14; First posted 2022-12-22 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Healthy
Keywords: Postmortem care; Creative drama; Nursing Students; Nursing Education

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled trial with experimental and control groups including pretest, posttest and persistence test.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessments will be performed by a investigator who was blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Creative Darama Group (Experimental): Postmortem care content including "The concept of death", "Postmortem Care", "Postmortem Care" and "Postmortem Care Practices" will be given to the students in the Creative Darama group in six sessions consisting of the preparation/warm-up, animation and evaluation stages of creative drama.
  Interventions: Other: Creative Darama Group
- Classical Education Group (Active Comparator): Theoretical training titled "Post-Death Care" and "The Concept of Death", "Post-Death Changes", "Post-Death Care" and "Post-Death Care Practices" will be conveyed to the students in the classical education group by the researcher using the method of direct expression. After the theoretical training, the students will be taken to the application laboratory and post-mortem care applications will be explained with the demonstration method.
  Interventions: Other: Classical Education Group

INTERVENTIONS:
Other: Creative Darama Group — Postmortem care training given by creative drama method
  Arms: Creative Darama Group
Other: Classical Education Group — Postmortem care training given by classical education method
  Arms: Classical Education Group

SUMMARY:
The goal of this randomized controlled including pretest, posttest and persistence test study is to examine the effect of creative drama method on student nurses' knowledge and skill levels related to postmortem care, learning permanence and satisfaction with the training method.

The main question it aims to answer are:

•Is the postmortem care training given to nursing students with the creative drama method effective on the level of knowledge and skills, the permanence of knowledge and skills and satisfaction with the training method? Participants will participate in an educational activity related to postmortem care. Researchers will compare it with the classical education method to see if postmortem care training given to nursing students with the creative drama method is effective.

DETAILED DESCRIPTION:
The research will be carried out in the form of determining the preliminary knowledge of nursing third year students about postmortem care, providing education with classical education and creative drama methods, evaluating the educational outcomes and permanence in education for knowledge and skills, and determining their satisfaction with the educational methods.

Hypotheses of the research are as follows. H1: There is a difference between the knowledge scores of the experimental and control groups on postmortem care. Is there a difference between the creative drama method and classical education method and the satisfaction of postmortem care students with the training method? H2: There is a difference between the skill scores of the experimental and control groups for postmortem care. H

: There is a difference between the information persistence scores of the experimental and control groups related to postmortem care.

H4: There is a difference between the skill persistence scores of the experimental and control groups for postmortem care.

H5: There is a difference between the satisfaction of the experimental and control groups with the training method

ELIGIBILITY:
Inclusion Criteria:

* Bolu Abant İzzet Baysal University Faculty of Health Sciences, Department of Nursing, 2022-2023 academic year fall semester to be studying in the third year.
* To have taken the "Principles of Nursing" course and the Loss-Death-Mourning process described in this context at the theoretical level.
* Agreeing to participate in the research.

Exclusion Criteria:

* Have previously received skills training related to postmortem care.
* Have previous clinical experience with postmortem care.
* Have previously provided postmortem care.
* Not agreeing to participate in the research.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2022-11-04 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Nursing students' level of knowledge about postmortem care:Pre-test | Just before training
  "Postmortem Care Knowledge Test" A "Postmortem Care Knowledge Test" consisting of 19 multiple-choice questions with five options has been developed to measure the level of knowledge of students on the subject of postmortem care. In the knowledge test, each question is 1 point. The score that can be obtained from the test varies between 0-19. The response time of the test is about 20 minutes. A high score from the test indicates that the level of postmortem care information is high, and a low level of postmortem care information is low.
Skill levels of nursing students in postmortem care:First-test | Immediately after training
  "Postmortem Care Skill Checklist" Postmortem Care Skill Checklist is a list of 25 items prepared by the researcher by using the process steps of postmortem care applications in the literature. The measurement criteria were prepared in the style of 3 likert as applied (2 points), partially applied (1 point) and did not apply (0 points). Each application item will be evaluated by averaging the scores given by two independent observers. The score that can be obtained from the applications is between 0-50. A high score obtained at the end of the evaluation indicates that the postmortem care skill level is high and the low postmortem care skill level is low.
Satisfaction levels of nursing students with the training method | Immediately after training
  "Satisfaction with Educational Methods Survey" "Satisfaction with Educational Methods Survey" is a questionnaire developed by Gürpınar and consists of 16 propositions (Cronbach alpha: 0.84). Each proposition is scored on a scale of 1 to 5 according to the 5-point lique. In the survey, at least 16 and at most 80 points are given to the satisfaction of the students from the educational methods It is determined that the satisfaction levels of the students increase as the score obtained from the survey increases, and the satisfaction levels decrease as they decrease

SECONDARY OUTCOMES:
Nursing students' level of knowledge about postmortem care:Post-test | Immediately after training
  "Postmortem Care Knowledge Test" A "Postmortem Care Knowledge Test" consisting of 19 multiple-choice questions with five options has been developed to measure the level of knowledge of students on the subject of postmortem care. In the knowledge test, each question is 1 point. The score that can be obtained from the test varies between 0-19. The response time of the test is about 20 minutes. A high score from the test indicates that the level of postmortem care information is high, and a low level of postmortem care information is low.

OTHER OUTCOMES:
Nursing students' level of knowledge about postmortem care:Persistence test | Four weeks after training
  "Postmortem Care Knowledge Test" A "Postmortem Care Knowledge Test" consisting of 19 multiple-choice questions with five options has been developed to measure the level of knowledge of students on the subject of postmortem care. In the knowledge test, each question is 1 point. The score that can be obtained from the test varies between 0-19. The response time of the test is about 20 minutes. A high score from the test indicates that the level of postmortem care information is high, and a low level of postmortem care information is low.
Skill levels of nursing students in postmortem care:Persistence test | Four weeks after training
  "Postmortem Care Skill Checklist" Postmortem Care Skill Checklist is a list of 25 items prepared by the researcher by using the process steps of postmortem care applications in the literature. The measurement criteria were prepared in the style of 3 likert as applied (2 points), partially applied (1 point) and did not apply (0 points). Each application item will be evaluated by averaging the scores given by two independent observers. The score that can be obtained from the applications is between 0-50. A high score obtained at the end of the evaluation indicates that the postmortem care skill level is high and the low postmortem care skill level is low.

CONTACTS AND LOCATIONS:
Overall Officials: Lütfiye Nur Uzun, PhD Student, Principal Investigator — Bolu Abant İzzet Baysal University Faculty of Health Sciences Nursing Department
Locations (1):
- Bolu Abant İzzet Baysal University Faculty of Health Sciences Nursing Department, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This study is planned as a doctoral thesis.